CLINICAL TRIAL: NCT01347320
Title: Clinical Impact of MR Imaging in Patients With Prostate Cancer
Brief Title: Preoperative Magnetic Resonance (MR) Imaging of Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Erik Rud, MD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OsloUH
Record Dates: First submitted 2010-03-09; First posted 2011-05-04 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; preoperative staging; MRI; Free surgical margins
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No preoperative MRI (No Intervention): control arm of the study
- MRI group (Active Comparator): preoperative MRI
  Interventions: Other: Preoperative MRI

INTERVENTIONS:
Other: Preoperative MRI — Preoperative staging
  Arms: MRI group

SUMMARY:
The investigators want to evaluate if preoperative MRI improves the surgical results, especially in respect to surgical margins. The impact on the surgical procedure will be evaluated.

In addition the investigators will examine the accuracy of tumor detection, localization and staging.

DETAILED DESCRIPTION:
Background:

During the last two decades, Magnetic Resonance Imaging (MRI) of the prostate has evolved to become a promising tool in preoperative evaluation of prostate cancer. Several studies have evaluated the radiological and histopathological correlation. However, the sensitivity and specificity in regard to staging have shown wide ranges and poor reproducibility. These discrepancies can be explained by difference in patient selection, MRI methods, and criteria used for diagnosis. More studies are therefore needed to evaluate the clinical impact of preoperative MRI in patients with prostate cancer.

Aims of the study:

To evaluate 1) detection rate of tumor 1-3 (tumor 1 = index tumor), size of tumor 1-3, possible extraprostatic extension and predict presence of Gleason grade 4 and 5 tumor, 2) the influence of preoperative MRI on the surgical decision process with respect to the operative procedure for removal of the gland and pelvic lymph node dissection, and 3) the impact of preoperative MRI on the rate of positive surgical margins and functional results.

Material and method:

A prospective study including 400 consecutive patients referred to robot assisted laparoscopic prostatectomy randomised to preoperative MRI (intervention group) and no MRI (control group). The prostatectomy specimens will be histopathologically examined, and TNM classification will be performed according to 2002 AJCC standard.

ELIGIBILITY:
Inclusion criteria

* All patients suitable for surgery.
* Positive biopsy (Gleason grade >3).
* Informed consent.

Exclusion Criteria:

* Patients who do not sign the consent paper for any reason or do not accept the study premises.
* Patents who want to withdraw for any reason during the study.
* Patients with contraindications to MRI (pacemaker, claustrophobia etc) and/or surgery.
* Patients who have undergone a high quality MRI examination of the prostate at another radiological center. In this situation the MR examination is evaluated together with the surgeon but the patient is not included in the study. (In case of a low quality examinations, we will disregard the findings, and include the patient).
* If the surgeon finds it unacceptable to perform RALP without MRI, because of various reasons (eg. patient demand, too high risk etc) the patient will not be included in the study.
* If preoperative MRI reveals extensive tumor invasion into adjacent organ (T4) or skeletal metastases (M1), as these cancer stadiums do not benefit from RALP.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2009-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Surgical margins | 30 days
  The surgical margins are assessed by evaluating the pathological specimen

SECONDARY OUTCOMES:
Surgical decision process | 30 days
  Evaluated using questionaire
Preoperative TNM classification | 1-4 weeks
  Based upon preoperative MRI
Detection of Gleason grade 4 and 5 | 30 days
Functional outcome | 1 year after prostatectomy
  Evaluate the functional outcome in respect to erectile dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Rud, MD, Principal Investigator — Oslo University Hospital, Aker
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Rud E, Baco E, Klotz D, Rennesund K, Svindland A, Berge V, Lundeby E, Wessel N, Hoff JR, Berg RE, Diep L, Eggesbo HB, Eri LM. Does preoperative magnetic resonance imaging reduce the rate of positive surgical margins at radical prostatectomy in a randomised clinical trial? Eur Urol. 2015 Sep;68(3):487-96. doi: 10.1016/j.eururo.2015.02.039. Epub 2015 Mar 23. PMID 25813692
- [Derived] Rud E, Klotz D, Rennesund K, Baco E, Johansen TE, Diep LM, Svindland A, Eri LM, Eggesbo HB. Preoperative magnetic resonance imaging for detecting uni- and bilateral extraprostatic disease in patients with prostate cancer. World J Urol. 2015 Jul;33(7):1015-21. doi: 10.1007/s00345-014-1362-x. Epub 2014 Jul 25. PMID 25059766